CLINICAL TRIAL: NCT02307981
Title: Management and Outcome of Visual Field Defects in Occipital Infarction (NOR-OCCIP)- A Multi-center Prospective Study
Brief Title: Norwegian Occipital Ischemic Stroke Study
Acronym: NOR-OCCIP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Stavanger HF (Other Government); St. Olavs Hospital (Other); Statped Vest (Unknown); Stavanger Municipality (Unknown)
Responsible Party: Principal Investigator, Kristin Modalsli Sand, Kristin Modalsli Sand MD, Haukeland University Hospital
Other Study IDs: 2012/2307
Record Dates: First submitted 2014-11-28; First posted 2014-12-04 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Ischemic Stroke; Visual Field Defect
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Visual field defect with vision teacher: Patients With occipital ischemic stroke and Visual Field defect that live in a geographical region where training With vision teacher is an available service (vision Teachers are a Limited Resource in Norway)
  Interventions: Other: Training with vision teacher (visual rehabilitation)
- Visual field defect without vision teacher: Patients With occipital ischemic stroke and a Visual Field defect, who live in a geographical area where training With vision teacher is not an available service.

INTERVENTIONS:
Other: Training with vision teacher (visual rehabilitation) — Individually adapted training With vision teacher
  Groups: Visual field defect with vision teacher

SUMMARY:
Patients who suffer an ischemic stroke in the occipital lobe often experience Visual Field defects. Visual Field defects are negatively correlated to falling, institutionalisation, rehabilitation outcome and quality of life. Patients are often not properly examined and seldom receive rehabilitation. NOR-OCCIP aims to evaluate the Natural history of Visual Field defects after occipital infarction and to determine whether rehabilitation is effective.

DETAILED DESCRIPTION:
BACKGROUND: Visual Field defects after cerebral infarction is an increasingly acknowledged problem, which has consequences for patient outcome. The aim of the Norwegian Occipital Ischemic Stroke Study (NOR-OCCIP) is to: 1.) Improve clinical diagnostics and management of visual field defects in occipital stroke. 2.) Identify and estimate the need for visual rehabilitation among patients with VFD by studying the natural course and the rate of spontaneous recovery. 3.) Study the effect of visual rehabilitation both on visual function as well as on quality of life. METHODS: Patients with acute ischemic occipital stroke on MRI are recruited from Bergen, Stavanger and Trondheim. Patients are included for a period of 1.5 years, starting August 15th 2013. Patients are eligible for inclusion if >18 years, written consent is obtained and the patient is able to co-operate to examination with autoperimetry. Within one week patients are examined by ophthalmologist after a standardized protocol including autoperimetry. During week four patients are examined by vision teacher after a standardized protocol and a structured interview on vision specific function and quality of life (VFQ-25) is conducted by a study nurse via telephone. If visual rehabilitation is provided by the municipality in which the patient lives, the patient will be referred to such. Eye examination including autoperimetry, vision teacher assessment and VFQ-25 is repeated after 6 months. All patients will be registered in the national stroke registry, and the following variables will be analysed: Demographic variables, lifestyle factors, clinical status at admission (scores on NIHSS), clinical status at discharge and 3 months post-stroke (scores on modified Rankin Scale). So far 62 patients have been included. Limited research exists on visual impairment after cerebral infarction. It is important to establish the natural course of visual impairment after ischemic stroke, and to evaluate the effect of visual rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Written consent obtained,
* age >18,
* acute occipital infarction on brain imaging and ability to cooperate for examination with autoperimetry

Exclusion Criteria:

* Pathological processes that severely affect eyesight.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital based
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-09 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Visual Field defect | 6 months
  Change in Visual Field defect as measured by autoperimetry

SECONDARY OUTCOMES:
Change in Visual function | 6 months
  Change in Visual function as measured by standardized mapping by vision teacher according to pre-specified protocol
Quality of life and self reported Visual function | 6 months
  Vision specific QoL and function as measured by VFQ-25
NIHSS | One week

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Modalsli Sand, MD, Principal Investigator — Haukeland University Hospital
Locations (2):
- Norway (2):
  - Stavanger University Hospital, Stavanger, Rogaland
  - St. Olav University Hospital, Trondheim